CLINICAL TRIAL: NCT01303978
Title: Open-label, Ascending-dose, Phase II Study to Determine the Minimum Effective Dose of APD421 in the Prevention of Cisplatin-induced Nausea and Vomiting
Brief Title: Phase II Proof-of-concept Study of APD421
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acacia Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DN10007
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- APD421 starting dose (Experimental)
  Interventions: Drug: APD421

INTERVENTIONS:
Drug: APD421 — Single dose

SUMMARY:
Evaluation of efficacy of APD421 in preventing nausea and vomiting caused by cisplatin

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age
2. Ability and willingness to give written informed consent
3. Patients scheduled to receive, on day 1 of their chemotherapy, a first cisplatin chemotherapy infusion at a dose of 50 mg/m2 or greater
4. Karnofsky performance score ≥ 60%
5. Adequate cardiac, hepatic and renal function

   * QTc interval < 500 ms
   * Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) < 5 x upper limit normal (ULN)
   * Bilirubin < 3 x ULN
   * Creatinine < 2 x ULN
6. Adequate haematological function

   * Haemoglobin ≥ 9 g/dL
   * White blood count ≥ 3.0 x 109/L
   * Platelet count ≥ 100 x 109/L
7. For females of child-bearing potential: ability and willingness to use a highly effective form of contraception (e.g., abstinence from sexual intercourse, surgical sterilisation (of subject or partner) or a double-barrier method of contraception such as either an intra-uterine device (IUD) or an occlusive cap with spermicide, in conjunction with partner's use of a condom) during the study and for a period of at least 48 hours afterwards.

Exclusion Criteria:

1. Patients scheduled to receive, prior to or in the 24 hours after cisplatin, any chemotherapeutic agent with a high or moderate emetic risk, see Appendix 4.
2. Patients scheduled to receive paclitaxel or docetaxel
3. Patients undergoing abdominal or pelvic irradiation within 48 hours prior to screening or scheduled to receive abdominal or pelvic irradiation between screening and 24 hours after cisplatin administration
4. Patients receiving APD421 for any indication within the last 2 weeks
5. Patients who are allergic to APD421 or any of the excipients of APD421
6. Patients with a pre-existing vestibular disorder
7. Patients being treated with regular anti-emetic therapy including corticosteroids
8. Patients receiving inhaled corticosteroids, unless started more than one month prior to the expected date of study entry
9. Patients being treated with medications which could induce torsades de pointes, including Class Ia antiarrhythmic agents such as quinidine, disopyramide, procainamide; Class III antiarrhythmic agents such as amiodarone and sotalol; and other medications such as bepridil, cisapride, thioridazine, methadone, IV erythromycin, IV vincamine, halofantrine, pentamidine, sparfloxacin
10. Patients being treated with xxx
11. Patients receiving benzodiazepines, unless on a stable dose for at least one month prior to the expected date of study entry
12. Patients with pre-existing nausea or vomiting in the 24 hours before receiving cisplatin chemotherapy, e.g. anticipatory emesis
13. Patients who are pregnant or breast feeding
14. Patients with a history of alcohol abuse
15. Patients with pre-existing, clinically significant cardiac arrhythmia
16. Any other concurrent disease or illness that, in the opinion of the investigator makes the patient unsuitable for the study
17. Patients who have participated in another study within the previous 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Complete Response | 24 hours after cisplatin dosing
  No emesis or use of rescue medication

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (3):
  - Herlev Hospital, Copenhagen
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- University Hospital of South Manchester NHS Trust, Manchester, United Kingdom